CLINICAL TRIAL: NCT07224191
Title: Human Hippocampal Oscillations During Visuomotor Exploration
Brief Title: Hippocampal Oscillations During Exploration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 25-01119; R61DC022830-01 (NIH)
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Epilepsy Surgery Patients (Experimental): Aim 1: Participants will be presented with between 10-15 unique immersive virtual environments (depending on patient tolerance) for patients to explore using VR glasses. Control tasks will be run to account for eye movements during non-navigation. For recording eye movements in darkness during REM sleep, as part of a control task, 4 electrodes will be placed above and below both eyes, a standard technique in polysomnographic studies.
  Interventions: Other: Visual Exploration
- Patients with RNS Devices (Experimental): Aim 2: Participants will walk between 4-6 rooms within an office floor. Each office will contain generic objects (office furniture, computers, lighting) and unique objects (artwork, photographs, books, and personal items). As control conditions, subjects will first be asked to walk around and between two empty rooms under different lighting conditions and speeds. Participants will also be asked to participate in all awake saccade control conditions (without a visual cognitive load).
  Interventions: Other: Ambulatory Exploration
- Healthy Control Participants (Experimental): Aim 2: Participants will walk between 4-6 rooms within an office floor. Each office will contain generic objects (office furniture, computers, lighting) and unique objects (artwork, photographs, books, and personal items). As control conditions, subjects will first be asked to walk around and between two empty rooms under different lighting conditions and speeds. Participants will also be asked to participate in all awake saccade control conditions (without a visual cognitive load).
  Interventions: Other: Ambulatory Exploration

INTERVENTIONS:
Other: Visual Exploration — Cognitive testing while admitted to the epilepsy monitoring unit (number of sessions will vary depending on patient availability and stamina).
  Arms: Epilepsy Surgery Patients
Other: Ambulatory Exploration — Series of cognitive tasks completed during a study visit.
  Arms: Healthy Control Participants; Patients with RNS Devices

SUMMARY:
The objective of this study is to determine how visuomotor exploration relates to hippocampal activity along its long axis. The study will investigate the neurophysiological mechanisms in the hippocampus during (1) visual exploration in surgical patients using high-resolution iEEG, and (2) ambulatory exploration in patients implanted with RNS devices.

DETAILED DESCRIPTION:
Aim 1 - Visual Exploration in Surgical Patients Investigators will study 20 surgical patients with high-resolution intracranial EEG (iEEG) to investigate hippocampal activity during visual exploration. Participants will view between 10-15 panoramic environments using Meta Quest AR/VR glasses while their eye movements and head turns are tracked. Eye-tracking, head-turn, and iEEG data will be synchronized with visual stimuli, and intracranial EEG and single-unit data will be analyzed for changes in neuronal firing and brain activity before and after saccades.

Aim 2 - Ambulatory Exploration in RNS Patients and Healthy Controls Investigators will study 12 epilepsy patients with implanted responsive neurostimulator (RNS) devices and 24 healthy controls (HCs) during real-world exploration. Participants will walk through and explore visually distinct rooms while wearing synchronized high-density EEG (hdEEG), eye-tracking glasses, and body position sensors. Data from hippocampal iEEG, hdEEG, eye tracking, and motion sensors will be synchronized offline to examine brain-behavior relationships and the influence of cognitive load on saccade-hippocampal interactions.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Adults (18-70 years)
* Able to provide informed consent

Aim 1: Surgical epilepsy patients' inclusion criteria

* Implanted hippocampal depth electrodes for Stage 1 epilepsy surgery
* IQ=>80*

Aim 2: RNS patients Inclusion criteria

* Implanted RNS device with at least one hippocampal depth electrode
* At least 5 months post-implantation to avoid the post-implant effect
* Have a relatively low number of seizures, defined as =<1 debilitating seizure per week
* Able to walk and wear research equipment without assistance
* IQ>=80

Aim 2: Healthy Control Inclusion criteria • Able to walk and wear research equipment without assistance

Exclusion Criteria:

RNS patients, Aim 2:

• Any generalized tonic-clonic seizure(s) within the last year

All subjects:

* Legally blind
* Smoking tobacco, marijuana, recreational drugs or alcohol use within 1 week of cognitive testing
* Unable to give informed consent
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-10-08 (Estimated); Study Completion 2028-10-08 (Estimated)

PRIMARY OUTCOMES:
Hippocampal Theta Power Under High Cognitive Loads | Study Visit (Day 1)
  Aims 1 and 2. High cognitive loads defined as visual exploration of a complex scene with goal-driven task.
Hippocampal Theta Power Under Medium Cognitive Loads | Study Visit (Day 1)
  Aims 1 and 2. Medium cognitive loads defined as visual exploration of a simpler scene with fewer objects.
Hippocampal Theta Power Under Low Cognitive Loads | Study Visit (Day 1)
  Aims 1 and 2. Low cognitive loads defined as visual exploration of moving dots.
Hippocampal Theta Power Under No Cognitive Loads | Study Visit (Day 1)
  Aims 1 and 2. Low cognitive loads defined as staring at a blank field of view or REM sleep.
Coherence Time-Locked to the Saccade Under High Cognitive Loads | Study Visit (Day 1)
  Aims 1 and 2. High cognitive loads defined as visual exploration of a complex scene with goal-driven task.
Coherence Time-Locked to the Saccade Under Medium Cognitive Loads | Study Visit (Day 1)
  Aims 1 and 2. Medium cognitive loads defined as visual exploration of a simpler scene with fewer objects.
Coherence Time-Locked to the Saccade Under Low Cognitive Loads | Study Visit (Day 1)
  Aims 1 and 2. Low cognitive loads defined as staring at a blank field of view or REM sleep.
Coherence Time-Locked to the Saccade Under No Cognitive Loads | Study Visit (Day 1)
  Aims 1 and 2. Low cognitive loads defined as staring at a blank field of view or REM sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Anli Liu, MD, MA, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The study will upload data into openneuro.org or comparable neuroscience data sharing platform, with data uploaded on a basis as specified by the conditions of awards supporting this research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to anli.liu@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.